CLINICAL TRIAL: NCT04196153
Title: A Comparison of Pedicle Screws Placement Accuracy in Thoracolumbar Spine Using Two Guidance Techniques: O-arm Navigation and Cervical Distractor Screws
Brief Title: Pedicle Screws Placement Accuracy in Thoracolumbar Spine Using O-arm Navigation VS Standard Cervical Distractor Screws
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kashabmo
Record Dates: First submitted 2019-12-07; First posted 2019-12-12 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Pedicle Screws; Surgery, Computer-Assisted/Adverse Effects; Bone Screws; Imaging, Three-Dimensional/Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuronavigation / O-arm group (Active Comparator): Under neural navigation with the use of intraoperative three dimensional imaging quality O-arm , pedicle screws inserted at the thoraolumbar/lumbar spine after insertion of the reference frame at the spinous process above or below the level of instrumentation followed by O-Arm imaging and uploading the images to the stelth navigation system and pedicle tract identification using instrumented tools guided by the Navigation polyaxial screws is inserted.
  Interventions: Procedure: Pedicle screws instrumentation
- Cervical distractor screws group (Active Comparator): pedicle screws inserted using marker screws after posterior exposure of thoracolumbar /lumbar spine by either open midline posterior exposure or minimal invasive posterior wiltse style exposure with expandable tubular retractor, anatomical landmark for insertion of pedical screws identified and followed by inserting of a cervical distraction screw size 3 / 12 mm as a stable marker using high speed drill. C-arm floro is used to take antroposterior and lateral view to confirm the position of the marker screws at this stage.free hand technique supported by the images provided to cannulate the pedicle with the use of information on the images taken for all the marker screws simultaneously.
  Interventions: Procedure: Pedicle screws instrumentation

INTERVENTIONS:
Procedure: Pedicle screws instrumentation — The screws are inserted in two or more consecutive levels to prevent motion at the segments that are being fused. It will be done using one of the two guidance technique depending on which arm the patient will be randomized to.

SUMMARY:
Pedicle screw instrumentation is used nowadays mostly in spine fusion which is a surgical option for treating variety of conditions such as vertebral fractures, degenerative spine diseases, spine tumors and spine deformities. However, pedicle screws misplacement and breach may occur and be a great cause of morbidity. The breach rate can be as high as 20-39.8% but most of the time only small number is associated with complications. Surgeons use assistive technique to avoid screw breached and improve screw placement accuracy. Investigators aim in this study to compare accuracy of pedicle screws placement using two guidance techniques are O-arm navigation the latest assistive imaging technique that uses three-dimensional (3-D) real time images to allow the surgeons follow the screw's trajectory, and standard cervical distractor screws to mark the entry point and trajectory.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need a thoracolumbar spine surgery that require pedicle screw insertion.

Exclusion Criteria:

* Patients whose surgeries in cervical spine
* Patients whose surgeries are for correction of deformities such as scoliosis and kyphosis, patients with infections or tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Rate screws breach | 6 months
  Investigators will determine the rate of screws breach in the two comparison groups
Screw insertion time | 5 hours
  screw insertion time in each technique which will be assessed by calculating the total time from puncture at the entry point by awl to complete all screw insertions into pedicles divided by the number of pedicle screws
screws revision times | 6 months
  investigators will determine which group needs more screws revision
degree of screws breach | 6 months
  Investigators will determine degree of screws breach in the two comparison groups

SECONDARY OUTCOMES:
Direction of the breach | 6 months
  investigators will ascertain direction of the breach, if it is lateral ,medial , inferior , or superior.
complications | Up to 24 weeks
  the two groups will be compared in rate of neurological or vascular complications.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Khashab, MD, Principal Investigator — Assistant Professor of Orthopedic, College of Medicine, KSAU-HS
Locations (1):
- King Abdulaziz Medical City, Jeddah, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] BOUCHER HH. A method of spinal fusion. J Bone Joint Surg Br. 1959 May;41-B(2):248-59. doi: 10.1302/0301-620X.41B2.248. No abstract available. PMID 13641310
- [Background] Gaines RW Jr. The use of pedicle-screw internal fixation for the operative treatment of spinal disorders. J Bone Joint Surg Am. 2000 Oct;82(10):1458-76. doi: 10.2106/00004623-200010000-00013. PMID 11057475
- [Background] Liljenqvist UR, Halm HF, Link TM. Pedicle screw instrumentation of the thoracic spine in idiopathic scoliosis. Spine (Phila Pa 1976). 1997 Oct 1;22(19):2239-45. doi: 10.1097/00007632-199710010-00008. PMID 9346144
- [Background] Krag MH, Beynnon BD, Pope MH, DeCoster TA. Depth of insertion of transpedicular vertebral screws into human vertebrae: effect upon screw-vertebra interface strength. J Spinal Disord. 1988;1(4):287-94. doi: 10.1097/00002517-198800140-00002. PMID 2980257
- [Background] Roy-Camille R, Saillant G, Mazel C. Internal fixation of the lumbar spine with pedicle screw plating. Clin Orthop Relat Res. 1986 Feb;(203):7-17. PMID 3955999
- [Background] Broom MJ, Banta JV, Renshaw TS. Spinal fusion augmented by luque-rod segmental instrumentation for neuromuscular scoliosis. J Bone Joint Surg Am. 1989 Jan;71(1):32-44. PMID 2913001
- [Background] Puvanesarajah V, Liauw JA, Lo SF, Lina IA, Witham TF. Techniques and accuracy of thoracolumbar pedicle screw placement. World J Orthop. 2014 Apr 18;5(2):112-23. doi: 10.5312/wjo.v5.i2.112. eCollection 2014 Apr 18. PMID 24829874
- [Background] Vaccaro AR, Rizzolo SJ, Balderston RA, Allardyce TJ, Garfin SR, Dolinskas C, An HS. Placement of pedicle screws in the thoracic spine. Part II: An anatomical and radiographic assessment. J Bone Joint Surg Am. 1995 Aug;77(8):1200-6. doi: 10.2106/00004623-199508000-00009. PMID 7642665
- [Background] Verma R, Krishan S, Haendlmayer K, Mohsen A. Functional outcome of computer-assisted spinal pedicle screw placement: a systematic review and meta-analysis of 23 studies including 5,992 pedicle screws. Eur Spine J. 2010 Mar;19(3):370-5. doi: 10.1007/s00586-009-1258-4. Epub 2010 Jan 6. PMID 20052504
- [Background] Gertzbein SD, Robbins SE. Accuracy of pedicular screw placement in vivo. Spine (Phila Pa 1976). 1990 Jan;15(1):11-4. doi: 10.1097/00007632-199001000-00004. PMID 2326693
- [Background] Kim TT, Drazin D, Shweikeh F, Pashman R, Johnson JP. Clinical and radiographic outcomes of minimally invasive percutaneous pedicle screw placement with intraoperative CT (O-arm) image guidance navigation. Neurosurg Focus. 2014 Mar;36(3):E1. doi: 10.3171/2014.1.FOCUS13531. PMID 24580001
- [Background] Luo TD, Polly DW Jr, Ledonio CG, Wetjen NM, Larson AN. Accuracy of Pedicle Screw Placement in Children 10 Years or Younger Using Navigation and Intraoperative CT. Clin Spine Surg. 2016 Apr;29(3):E135-8. doi: 10.1097/BSD.0000000000000230. PMID 27007788
- [Background] Scarone P, Vincenzo G, Distefano D, Del Grande F, Cianfoni A, Presilla S, Reinert M. Use of the Airo mobile intraoperative CT system versus the O-arm for transpedicular screw fixation in the thoracic and lumbar spine: a retrospective cohort study of 263 patients. J Neurosurg Spine. 2018 Oct;29(4):397-406. doi: 10.3171/2018.1.SPINE17927. Epub 2018 Jul 6. PMID 29979141
- [Background] Tajsic T, Patel K, Farmer R, Mannion RJ, Trivedi RA. Spinal navigation for minimally invasive thoracic and lumbosacral spine fixation: implications for radiation exposure, operative time, and accuracy of pedicle screw placement. Eur Spine J. 2018 Aug;27(8):1918-1924. doi: 10.1007/s00586-018-5587-z. Epub 2018 Apr 17. PMID 29667139